CLINICAL TRIAL: NCT06218121
Title: Update on the Detection of Frailty in Older Adults: A Multicenter Cohort Machine Learning-Based Study
Brief Title: Update on the Detection of Frailty in Older Adults
Status: Recruiting | Type: Observational
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Principal Investigator, Eleuterio Atanasio Sánchez Romero, Principal Investigator, Universidad Europea de Madrid
Other Study IDs: Detection of Frailty
Record Dates: First submitted 2024-01-02; First posted 2024-01-23 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Strength; Quality of Life; Functional Independence; Functionality; Pain; Sarcopenia; Anxiety; Kinesiophobia; Depression
Keywords: Frailty; Quality of life; Sarcopenia; Ultrasound
MeSH Terms: conditions — Pain; Sarcopenia; Anxiety Disorders; Kinesiophobia; Depression; Frailty | interventions — Nutritional Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Frail Older Adult Patients: For the cohort study, 500 frail older adult patients will be evaluated by means of instrumental and functional tests that assess their functional capacity, in addition to ultrasound imaging to study sarcopenia and nutrition, as well as psychological variables. The correlation between all functional, ultrasound, nutritional, and psychological variables will be analyzed. Through GLIM diagnosis, anthropometric data (weight, height, BMI) as well as analytical data including inflammation information (CRP and albumin) will be used to reach a diagnosis that allows comparison/correlation with the rest of the variable parameters. All available information will be collected during the follow-up in order to generate Machine Learning on the objective evolution and symptomatology of these patients, generating profiles that facilitate the most accurate and appropriate treatment for each patient.
  Interventions: Diagnostic Test: Instrumental and Functional Tests that Assess Functional Capacity

INTERVENTIONS:
Diagnostic Test: Instrumental and Functional Tests that Assess Functional Capacity — The correlation between all functional, ultrasound, nutritional, and psychological variables will be analyzed. Through GLIM diagnosis, anthropometric data (weight, height, BMI) as well as analytical data including inflammation information (CRP and albumin) will be used to reach a diagnosis that allows comparison/correlation with the rest of the variable parameters.
  Other Names: Ultrasound Imaging to Study Sarcopenia and Nutrition; Psychological Variables.

SUMMARY:
The main objective is to update the diagnostic assessment of frailty by correlating several variables with the ultrasound image of the frail elderly patient.

Secondarily, the investigators intend to collect and analyze data on functional capacity and quality of life variables on the evolution of musculoskeletal symptoms, as well as on pain and psychological variables. Similarly, it is intended to make a record of different profiles and subtypes of frail older adult patients to be stored in Machine Learning in order to establish therapeutic intervention plans that allow both the evaluation and treatment of patients.

DETAILED DESCRIPTION:
The present cohort study will be conducted in 500 older adults diagnosed with frailty.

The correlation of the demographic variables, physical functionality tests and psychoemotional constructs that will be analyzed in this study with the ultrasound image obtained from the patients will improve the ultrasound diagnosis of frailty, providing new information that will facilitate the work of healthcare personnel in the diagnosis and management of frailty.

Similarly, the use of Machine Learning will allow institutions to extract data on different patient profiles, signs and symptoms of frailty and the different risk factors that affect frailty patients, which will improve treatments and favor the development of educational programs tailored to the patient's needs.

ELIGIBILITY:
Inclusion Criteria:

A diagnosis of signs and symptoms of frailty by a geriatric physician in the research group will be used as the primary inclusion criterion. Frailty will be assessed and diagnosed using the frailty phenotype and the Clinical Frailty Scale.

Exclusion Criteria:

* Acute myocardial infarction in the last 3 months and/or unstable angina pectoris
* Uncontrolled arrhythmia, recent thromboembolism and terminal illness.
* Patients undergoing MMII unloading or MMSS/MMII fractures in the last three months.
* Patients with a functional gait index of 1 (Inability to walk)
* Severe pain (7/10 VAS)
* Previous neuromuscular pathology presenting with weakness
* Medication that does not allow the patient's actual muscle reaction to be assessed
* Severe cognitive impairment that would prevent collaboration and understanding of the tests to be performed.
* Cardiovascularly unstable patients and uncontrolled arterial hypertension.

Min Age: 62 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The present cohort study will be conducted in older adults diagnosed with frailty. A multicenter study will be conducted among the Residencia de Nuestra Señora de la Soledad y del Carmen (Colmenar Viejo, Madrid), Residencia San Camilo (Tres Cantos, Madrid), Centro de Día San Camilo (Tres Cantos, Madrid), Residencia San Luis de Gonzaga (Carretera de Colmenar Viejo), Hospital Universitario Rey Juan Carlos (Móstoles, Madrid) and Hospital Puerta de Hierro (Majadahonda, Madrid) from their diagnosis
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-04-20 (Actual); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Manual Grip Strength | Baseline
  The grip strength in both hands will be measured by measuring the maximum grip strength. A bulb dynamometer will be used for this measurement.
Quality of Life (EQ-5D-5L) | Baseline
  It will be evaluated by means of the the EuroQol 5-dimensions 5-levels (EQ-5D-5L), which is a generic instrument for measuring health-related quality of life. The patient himself assesses his state of health, in levels of severity by dimensions The first allows the respondent to define the state of health according to the EQ-5D multi-attribute classification system, composed of 5 dimensions (mobility, self-care, activities of daily living, pain/discomfort and anxiety/depression), and in each of them there are 3 levels of severity (1, 2 or 3).
Basic Activities in Daily Life | Baseline
  The Barthel Index evaluated one's ability to care for him/herself through ten activitiesof daily living like feeding, bathing, grooming, dressing, bowel and bladder control,toileting, chair transfer, ambulation, and stair climbing; the maximum score is 100 pointsand the higher the score, the greater the functional independence of the patient. Thefollowing baseline data regarding age, sex, and admission diagnosis were also collected .
Balance | Baseline
  The Trunk Control Test (TCT) evaluated four aspects of trunk movement, swinging to both sides, sitting balance, and rising from the floor; individual items are scored from 0 (incapable) to 12 (ability to perform the movement but with an unusual style) and 25 (ability to perform the movement correctly).
Visual Analog Scale (VAS) | Baseline
  To evaluate the pain that the patient has, we use the VAS. This is a 100 mm line that measures pain intensity. The left end of the line represents the absence of pain, while the right end represents the worst pain imaginable. The numerical pain intensity scale adds a numerical graduation where 1 is no pain and 10 is the worst pain imaginable. The confidence and reliability of this scale has been approved and validated in different studies.
Strength | Baseline
  The Medical Research Council Sum Score (MRCSS) strength assessment scale evaluated muscle strength in the upper and lower limbs. The different movements evaluated arescored from 0 to 5 and a maximum score of 60 can be obtained.
Anxiety | Baseline
  Anxiety was measured with Spanish version of State-trait Anxiety Inventory (STAI). Scores of 20-37 indicate no or low anxiety; 38-44 moderate anxiety; 45-80 high anxiety.
Kinesiophobia | Baseline
  Kinesiophobia was measured with Spanish version of Tampa Scale of Kinesiophobia. Higher scores denotes greater fear of experiencing pain while moving.
Depression | Baseline
  Depressive symptoms were measured with Spanish version of Beck Inventory II. 0-13 normal scores; 14-19 mild; 20-28 moderate; 29-63 severe depression.
Risk of Falls | Baseline
  Assessment of fall risk according to the Vivifrail protocol: cumulative number of falls in the past year, cumulative number of falls with physician care, suffer at least 1 fall in the past year, Timed Up and Go test (TUG) and existence of dementia to establish the existence of fall risk (+ or -); the TUG assesses the time it takes to get out of the chair, walk three meters, back to the chair, and to sit down.

CONTACTS AND LOCATIONS:
Overall Officials: Eleuterio A. A. Sánchez Romero, PhD, Principal Investigator — European University of Madrid
Locations (1):
- Hospital Puerta de Hierro de Majadahonda, Madrid, Outside of the US, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fernandez-Carnero S, Martinez-Pozas O, Pecos-Martin D, Pardo-Gomez A, Cuenca-Zaldivar JN, Sanchez-Romero EA. Update on the detection of frailty in older adults: a multicenter cohort machine learning-based study protocol. Aging (Albany NY). 2025 May 21;17(5):1328-1339. doi: 10.18632/aging.206254. Epub 2025 May 21. PMID 40413725